CLINICAL TRIAL: NCT03020875
Title: Single-Center, Randomized Controlled Trial of Intravenous v Oral Acetaminophen Administration in Perioperative Care of 1 and 2 Level XLIFs Supplemented With Bilateral Pedicle Screw Stabilization: a Comparative Effectiveness Study
Brief Title: IV vs Oral Acetaminophen in Spine Fusion Perioperative Care
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-516
Record Dates: First submitted 2016-07-05; First posted 2017-01-13 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2024-04

CONDITIONS: Multimodal Analgesic Approach
Keywords: Acetaminophen; Pain management
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- PO Acetaminophen (Active Comparator): Preop:
  Eligible patients will receive oral acetaminophen within 3 hours of OR start time.
  Postop:
  Eligible patients will be administered oral acetaminophen following 1 and 2 level LLIFs supplemented with instrumented posterior fusion to evaluate pain management outcomes. Dosing for the group will be the following:
  • Oral Acetaminophen 1,000 mg every 6 hours for 48 hours postoperative. Medication will be given at least 6 hours following initial preoperative dose of oral acetaminophen.
  Postop supplemental pain medications:
  All patients will receive a standardized hydromorphone IV-PCA order set for 24 hours postoperatively. The use of tramadol and tapentadol will specifically be discouraged due to challenges in determining morphine-equivalent dosing with these specific agents. Similarly, acetaminophen containing combination products (e.g. oxycodone/acetaminophen or hydrocodone/acetaminophen) will not be allowed due to overlap with the primary study medications.
  Interventions: Drug: Per Os Acetaminophen
- Intravenous Acetaminophen (Active Comparator): Preop:
  Eligible patients will receive IV acetaminophen within 3 hours of OR start time.
  Postop:
  Eligible patients will be administered IV acetaminophen following 1 and 2 level LLIFs supplemented with instrumented posterior fusion to evaluate pain management outcomes. Dosing for the group will be the following:
  • IV Acetaminophen 1,000 mg [100 ml] every 6 hours for 48 hours postoperative. Medication will be given at least 6 hours following initial preoperative dose of IV acetaminophen.
  Postop supplemental pain medications:
  All patients will receive a standardized hydromorphone IV-PCA order set for 24 hours postoperatively. The use of tramadol and tapentadol will specifically be discouraged due to challenges in determining morphine-equivalent dosing with these specific agents. Similarly, acetaminophen containing combination products (e.g. oxycodone/acetaminophen or hydrocodone/acetaminophen) will not be allowed due to overlap with the primary study medications.
  Interventions: Drug: Ofirmev

INTERVENTIONS:
Drug: Ofirmev — Intravenously administered acetaminophen.
  Other Names: Intravenous Acetaminophen
  Arms: Intravenous Acetaminophen
Drug: Per Os Acetaminophen — Orally administered acetaminophen.
  Arms: PO Acetaminophen

SUMMARY:
The United States is currently experiencing an explosive opioid epidemic. In 2014 alone, 28,647 Americans died from an opioid associated overdose; the annual death toll has increased by over 300% since 2000. The epidemic poses a complex scenario for physicians administering treatment for postoperative pain, as opioids are key analgesic agents in treating moderate to severe pain. In order to reduce the patients risk for long term opioid use and the associated side effects, physicians have begun shifting to multimodal analgesic approaches to treat postoperative pain. These approaches have been found to be similarly efficacious, while also reducing opioid usage and associated side effects, such as: nausea, vomiting, and ileus.

This study proposes a multimodal analgesic approach, which the investigators believe will reduce short and long term opioid usage, the associated side effects, and the financial burden. Intravenous acetaminophen is an effective medication for both primary and adjunctive pain management, however its use is limited by a high cost to perceived benefit ratio. Oral acetaminophen is a relatively inexpensive option, although perhaps less effective than the IV option, and also often not feasible to utilize in the immediate post-operative period when patients are unable to safely swallow pills. The hypothesis of this investigation is to understand if adding intravenous acetaminophen to the perioperative care regimen after lumbar spinal surgery will result in improved pain management in the perioperative period while decreasing opioid usage and related complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spinal stenosis of the lumbar spine with degenerative spondylolisthesis
* Skeletally mature adults between the ages of 18-85 years at the time of surgery
* The greater of the patients right and left VAS leg pain, or back pain, score is > 40 mm on a 100 mm scale
* Has attempted conservative therapy
* Psychosocially, mentally, and physically able to fully comply with this protocol, including adhering to scheduled visits, treatment plan, completing forms, and other study procedures
* Personally signed and dated informed consent document prior to any study-related procedures indicating that the patient has been informed of all pertinent aspects of the study

Exclusion Criteria:

* Any evidence of a prior/current fracture, compromised vertebra, current or past trauma, or tumor at affected level or the spinous processes at the adjacent levels
* Revision of prior fusion attempt at the level being operated on
* Cauda Equina Syndrome defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder dysfunction (bladder retention or incontinence)
* Significant peripheral neuropathy or acute denervation secondary to radiculopathy, caused by conditions other than spinal stenosis
* Significant peripheral vascular disease (diminished dornails pedis or tibial pulses)
* Morbid obesity, defined as BMI > 40 kg/m2; or underweight, defined as BMI < 18.5 kg/m2
* Active systematic or local infection
* Active Viral Hepatitis (receiving medical treatment within 1 year); or any other acute hepatitis within the past 6 months
* Immunocompromised such as but not limited to Acquired Immunodeficiency Syndrome (AIDS), HIV infection, Severe Combined Immunodeficiency Syndrome, Thymic Hypoplasia
* Insulin dependent diabetes mellitus or any other medical conditions that would represent a significant increase in surgical risk or interfere with normal healing
* Immunologically suppressed, or has received systemic steroids, excluding nasal steroids, at any dose for >1 month within last 12 months
* History of Paget's disease, osteomalacia, or osteoporosis with a DEXA t-score less than or equal to -2.5
* Active malignancy. A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and there has been no clinical signs or symptoms of the malignancy >5 years
* Any current history of substance abuse (e.g., recreational drugs, narcotics, or alcohol)
* History of psychosocial disorders that could prevent accurate completion of self-reporting assessment scales
* Previous known allergy to acetaminophen
* Women who are pregnant or lactating
* Patients involved in active litigation relating to his/her spinal condition
* Patients taking >30mg/day of oral morphine sulfate, or the equivalent of this daily for more than 3 months
* Patient is unable to ingest orally administered medication
* Patient receiving autologous Iliac Crest bone graft (ICBG)
* Known intolerance of or true allergy to hydromorphone or oxycodone.
* History of moderate to severe Cirrhosis, defined as Child Pugh score of class B, C, or D
* History of Hemochromatosis or Porphyria
* Patient taking Isoniazid or barbiturates

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2017-01; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for back and legs | Change from baseline VAS at 6 months postoperative
  Self reported pain frequency and intensity at 24 hour postoperative intervals until patient is discharged, at 6 week and 6 month follow-up. The scale is scored on a 100 mm line, with 0 being no pain and 100 being worst pain imaginable.

SECONDARY OUTCOMES:
Length of Stay (LOS) | Immediate postoperative
  Measured in total hours until discharge from hospital
Opioid Equivalent Dosing during Hospital Stay | Postoperative
  Measured every 24 hours postoperative until discharge from hospital
Time to Ambulation | Immediate postoperative
  Measured in total hours postoperative until patient is ambulatory
Oswestry Disability Index Version 2.1 (ODI) | Preoperative, 6 weeks and 6 months postoperative
Long Term Opioid Usage | 6 months Postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Chad Craig, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided